CLINICAL TRIAL: NCT06380907
Title: A Randomized, Double-Blind, Vehicle-Controlled, Multicenter, Dose-Ranging, Phase 2 Study to Evaluate the Efficacy and Safety of Different Doses of ZL-1102 Topical Gel (A Human VH IL-17A Antibody Fragment) in the Treatment of Chronic Plaque Psoriasis
Brief Title: A Phase 2 Study of ZL-1102 in Patients With Chronic Plaque Psoriasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zai Lab (Hong Kong), Ltd. (Industry)
Collaborators: Zai Lab (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZL-1102-002
Record Dates: First submitted 2022-11-15; First posted 2024-04-24 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Arm 1 (Active Comparator): ZL-1102
  Interventions: Drug: ZL-1102 1% w/w gel BID for 16 weeks
- Arm 2 (Active Comparator): ZL-1102
  Interventions: Drug: ZL-1102 3% w/w gel BID for 16 weeks
- Arm 3 (Active Comparator): ZL-1102
  Interventions: Drug: ZL-1102 3% w/w gel QD for 16 weeks
- Arm 4 (Placebo Comparator): Vehicle
  Interventions: Drug: Placebo ZL-1102 0% w/w gel BID for 16 weeks
- Arm 5 (Placebo Comparator): Vehicle
  Interventions: Drug: Placebo ZL-1102 0% w/w gel QD for 16 weeks

INTERVENTIONS:
Drug: ZL-1102 1% w/w gel BID for 16 weeks — ZL-1102
  1% w/w gel BID for 16 weeks
  Arms: Arm 1
Drug: ZL-1102 3% w/w gel BID for 16 weeks — ZL-1102 3% w/w gel BID for 16 weeks
  Arms: Arm 2
Drug: ZL-1102 3% w/w gel QD for 16 weeks — ZL-1102 3% w/w gel QD for 16 weeks
  Arms: Arm 3
Drug: Placebo ZL-1102 0% w/w gel BID for 16 weeks — Vehicle 0% w/w gel BID for 16 weeks
  Arms: Arm 4
Drug: Placebo ZL-1102 0% w/w gel QD for 16 weeks — Vehicle 0% w/w gel QD for 16 weeks
  Arms: Arm 5

SUMMARY:
A Randomized, Double-Blind, Vehicle-Controlled, Multicenter, Dose-Ranging, Phase 2 Study to Evaluate the Efficacy and Safety of Different Doses of ZL-1102 Topical gel (A Human VH IL-17A Antibody Fragment) in the Treatment of Chronic Plaque Psoriasis

DETAILED DESCRIPTION:
This is a randomized, double-blind, vehicle-controlled, dose-ranging, phase 2 study of ZL-1102 in patients with chronic plaque psoriasis. Approximately 250 patients will be randomized at a ratio of 1:1:1:1:1 to 5 treatment arms for 16 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age.
2. Willing and able to provide signed and dated informed consent prior to any study-related procedures, and willing and able to comply with all study procedures
3. Clinical diagnosis of psoriasis vulgaris of at least 6 months duration as determined by Investigator via medical records or in medical history obtained from the patient, is currently eligible for topical treatment and meets all the following criteria at screening and baseline:

   1. IGA ≥ 2 (5 score system)
   2. Affected BSA 3%-15% (excluding head)
4. Agree not to have prolonged sun exposure (e.g., recreational) during the study period. Tanning bed use or use of other light-emitting diodes (LEDs) is not allowed.

Exclusion Criteria:

1. Other types of psoriasis dominant other than plaque psoriasis (e.g., psoriatic arthritis, pustular, erythrodermic, guttate, palmar, plantar, scalp or nail disease) or the lesion is not eligible for topical treatment only.
2. Patients with any serious medical/psychiatric condition or clinically significant laboratory abnormality that would prevent study participation or place the patient at significant risk, as determined by the Investigator.
3. Known or suspected:

   1. Severe renal insufficiency or hepatic insufficiency.
   2. History of severe depression or suicidal ideation or behavior within 2 years prior to screening.
4. Positive for any of the following tests at screening:

   1. Human immunodeficiency virus (HIV): HIV antibody
   2. Hepatitis B virus (HBV): hepatitis B surface antigen (HBsAg)/hepatitis B core antibody (HBcAb)/HBV DNA
   3. Hepatitis C virus (HCV): HCV RNA
5. Patients with active tuberculosis (TB) or untreated latent TB per local guidelines.
6. History of and/or concurrent condition of inflammatory bowel disease (IBD) (ulcerative colitis and Crohn's disease), or signs/symptoms of IBD at screening that, in the opinion of the Investigator, pose an unacceptable risk to the patient if participating in the study.
7. History of and/or concurrent condition of serious hypersensitivity (anaphylactic shock or anaphylactoid reaction) to IL-17 antibodies and any human or humanized biological agents.
8. Patients who have a history of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥ 3 years before the initiation of study treatment.
9. Patients with a history of chronic alcohol or drug abuse within 6 months of the initiation of study treatment, as determined by the Investigator.
10. Prior exposure to ZL-1102.
11. Patients who have received a live vaccine within 6 weeks prior to dosing on Day 1.
12. Females who are pregnant, wishing to become pregnant during the study, or are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of different doses of ZL-1102 compared to Vehicle at Week 16. | 16 weeks
  The proportion of patients achieving mPASI 75 (at least a 75% reduction in mPASI score from baseline) at Week 16.

SECONDARY OUTCOMES:
The proportion of patients achieving IGA treatment success. | 20 Weeks
  The proportion of patients achieving IGA treatment success, defined as an IGA score of 0 or 1 with at least a 2-point improvement from baseline at Weeks 2, 4, 8, 12, 16,and 20.
The proportion of patients achieving IGA score of 0 or 1. | 20 Weeks
  The proportion of patients achieving an IGA score of 0 or 1 at Weeks 2, 4, 8, 12, 16, and 20
The percent change from baseline in mPASI score. | 20 Weeks
  The percent change from baseline in mPASI score at Weeks 2, 4, 8, 12, 16, and 20.
The proportion of patients achieving mPASI 75 at Week 2, 4, 8, 12, and 20. | 20 Weeks
  The proportion of patients achieving mPASI 75 at Week 2, 4, 8, 12, and 20.
The proportion of patients achieving mPASI 50/90/100 at Weeks 2, 4, 8, 12, 16, and 20. | 20 Weeks
  The proportion of patients achieving mPASII 50/90/100 at Weeks 2, 4, 8, 12,16, and 20.
Time to achieve mPASI 50/75/90. | 20 Weeks
  The time to achieve mPASI 50/75/90 through week 20.
Time to achieve IGA score of 0 or 1. | 20 Weeks
  Time to achieve IGA score of 0 or 1 through Week 20.
Time to achieve 1- or 2-point improvement in IGA. | 20 Weeks
  Time to achieve 1- or 2-point improvement in IGA score through Week 20.
Incidence of Treatment Related Adverse Events through Week 20. | 20 Weeks
  Number of patients with treatment related adverse events through week 20.
Mean local tolerability scores (LTS) | 20 Weeks
  Mean local tolerability scores at Weeks 2, 4,8, 12,16, and 20
Serum concentration of ZL-1102. | 16 Weeks
  Serum concentration of ZL-1102.
Anti-drug antibody (ADA) of ZL-1102. | 16 Weeks
  Incidence, prevalence, and titers of ADA of ZL-1102 in this study

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (10):
  - Zai Lab Site 5013, Phillip, Australian Capital Territory
  - Zai Lab Site 5021, Kogarah, New South Wales
  - Zai Lab Site 5016, Kotara, New South Wales
  - Zai Lab Site 5020, Birtinya, Queensland
  - Zai Lab Site 5019, Coorparoo, Queensland
  - Zai Lab Site 5017, Woolloongabba, Queensland
  - Zai Lab Site 5014, Carlton, Victoria
  - Zai Lab Site 5015, Melbourne, Victoria
  - Zai Lab Site 5002, Melbourne E., Victoria
  - Zai Lab Site 5018, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No